CLINICAL TRIAL: NCT01665456
Title: Assessing Childbirth-related Complications at the Community Level in Kenya: A Case Control Study Among Postpartum Women
Brief Title: Assessing Childbirth-related Complications at the Community Level in Kenya
Status: Completed | Type: Observational
Sponsor: Wilson Liambila (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Wilson Liambila, Senior Programme Officer, Kenyatta National Hospital
Organization: Kenyatta National Hospital (Other Government)
Other Study IDs: P141/03/2012
Record Dates: First submitted 2012-08-09; First posted 2012-08-15 (Estimated); Last update posted 2014-04-28 (Estimated); Status verified 2014-04

CONDITIONS: Puerperal Sepsis; Postpartum Hemorrhage; Preeclampsia and Eclampsia; Retained Placenta, Without Hemorrhage; Obstructed Labor Due to Breech Presentation
Keywords: complications
MeSH Terms: conditions — Puerperal Infection; Postpartum Hemorrhage; Pre-Eclampsia; Eclampsia; Placenta, Retained

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: None Retained — This was a two-arm study (Cases and controls). Random identification of cases through cross-sectional survey was done. Then, a random sample of controls was drawn from the source population from which the cases were selected (i.e. from same study base except that they were not cases) through matching variables i.e. age and location. Individual matching of controls to the characteristics of the cases was done. A total of 585 clients (women) were recruited (294cases and 291 controls).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cases (women with complications): Cases are women aged 15-49 years who delivered within 12 months prior to data collection and had experienced obstetric complication(s) that either necessitated treatment or hospitalization in order to prevent the likelihood of death of the mother.
- Control (women who did not experience any complications): Controls are women aged 15-49 years who delivered within 12 months prior to data collection. They did not have or develop any of the complications which cases experienced or suffered from.Although controls did not have complications, they were individually matched on the basis of age and location. The idea was to compare how many cases were exposed versus how many controls were exposed.

SUMMARY:
Kenya is one of the countries in sub-Saharan Africa that still experience high maternal mortality. For instance, in 2008/09 maternal mortality ratio was estimated to be 488/100,000 live births. Direct obstetric complications such as puerperal sepsis, postpartum hemorrhage, pre-eclampsia and eclampsia, obstructed labor and indirect causes including HIV, malaria and anemia in pregnancy are responsible for the majority of these cases. Just under 44% of births in Kenya are delivered under the supervision of a skilled birth attendant.

The overall objective of this study is to determine the effect of provider type in the occurrence and management of serious childbirth related complications among postpartum women at the community level in Bungoma and Lugari Districts of Western Province, Kenya.

The proposed study will employ a case control study design in which women with obstetric complication(s)will be cases and women without obstetric complications will be controls. Controls will be sampled concurrently with the cases. Each time a new case is diagnosed, a control is selected from the population at risk in the neighborhood at that point in time.

The study population will consist of women aged 15-49 years with a delivery in the past 12 months. A woman who reports having experienced a birth-related complication will be recruited as a case while woman who reports having experienced no complication during child-birth will be recruited as a control.

DETAILED DESCRIPTION:
Evidence from published literature is scanty on the effect of various categories of health providers in averting serious child birth related complications at the community level. For instance, no one knows what happens to pregnancy outcomes for both the mother and the baby in a context where a significant proportion of women are delivered by neighbors, relatives or on their own. Literature is also scanty regarding the outcomes of child birth related complications in situations where Traditional Birth Attendants conduct a significant proportion of deliveries.

A thorough understanding of factors that fuel disrespect and abuse as well as their effect on utilization of delivery services will help providers and programme managers to explore ways of addressing this issue. This study hypothesizes that since majority of deliveries take place at the household level, most complications and even deaths are likely to occur at this level.

The overall objective of this study is to determine the effect of provider type in the occurrence and management of serious childbirth related complications among postpartum women at the community level in Bungoma and Lugari Districts of Western Province, Kenya. Specific objectives of the study are:

To determine the quality of obstetric care given by community midwives and TBAs to clients seeking antenatal care, during delivery and post-partum care at the community level by assessing providers' preparedness and the range of services offered.

To assess the nature of obstetric complications among those women who were delivered by skilled health providers, versus those who were delivered by TBAs, neighbors, friends or on their own To determine the role of socio-economic, demographic and health service related factors in the occurrence of child birth related complications at the community level To obtain views from key stakeholders on the extent and occurrence of child birth related complications at the community level

ELIGIBILITY:
Case Inclusion criteria:

* Delivery in the past 12 months
* Suffered from obstetric complications during child birth and within 42days
* Provided oral or written informed consent to participate in the study
* Age ranges 15-49 years

Control inclusion criteria

* Delivered in the past 12 months
* Did not suffer from obstetric complications during child birth and within 42 days after delivery
* Provided oral or written informed consent to participate in the study
* Age ranges 15-49 years

Case and Control exclusion criteria:

* Did not deliver in the past 12 months;
* Refused to participate in the study;
* Excluded as controls if experienced complications similar to cases
* Excluded as cases if they didnot experience complications
* If unable to give informed consent or follow an interview

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population consisted of women aged 15-49 years with a delivery within 12 months preceding data collection date. A woman who reported having experienced a birth-related complication was recruited as a case. A woman aged 15-49 years with a delivery within 12 months preceding data collection who report having experienced no complication during child-birth was recruited as a control.
Sampling Method: Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2012-08; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
The odds ratio was the primary outcome measure of association between the the occurrence of complications and exposure to health providers in the past 12 months. | One Year
  The study sought to determine the association of provider type with the occurrence and management of serious childbirth related complications among postpartum women at the community level in Kenya in the past 12 months.The odds of exposure among cases were compared to the odds of exposure among controls to estimate the magnitude of association between exposure to health providers and other caregivers and the occurrence of complications.

SECONDARY OUTCOMES:
Proportion of women receiving skilled attendance at birth in the community in the past 12 months. | One Year
  This secondary outcome measure was assessed by collecting information on the nature of obstetric complications among those women who were delivered by skilled health providers, versus those who were delivered by Traditional Birth attendants, neighbours, friends or delivered on their own.

OTHER OUTCOMES:
Proportion of women with obstetric complications reporting to have been referred within 0-4 hours and 5-8 hours of admission or assessment to another level of care in the past 12 months. | One Year
  Prompt referral of women with obstetric complications is critical to their survival.Data was captured on the proportion of pregnant women in labour or in the postpartum period who were referred within 0-4hours and 5-8hours by health care providers or other care givers at the community level to the next level of care or the nearest health facilities after assessing or examining them.

CONTACTS AND LOCATIONS:
Overall Officials: Shiphrah N. Kuria, MB ChB, MMed (OBGYN), Principal Investigator — Division of Reproductive Health- Ministry of Public Health and Sanitation; Wilson N. Liambila, MSc, Principal Investigator — Population Council
Locations (1):
- Lugari and Bungoma districts, Kakamega, Western Province, Kenya

REFERENCES:
- [Background] Brennan M. Training traditional birth attendants reduces maternal mortality and morbidity. Trop J Obstet Gynaecol. 1988;1(1):44-7. PMID 12179276
- [Result] Koblinsky MA, Tinker A, Daly P. Programming for safe motherhood: a guide to action. Health Policy Plan. 1994 Sep;9(3):252-66. doi: 10.1093/heapol/9.3.252. PMID 10137741
- [Result] Bisika T. The effectiveness of the TBA programme in reducing maternal mortality and morbidity in Malawi. East Afr J Public Health. 2008 Aug;5(2):103-10. PMID 19024419
- [Result] Magoma M, Requejo J, Campbell OM, Cousens S, Filippi V. High ANC coverage and low skilled attendance in a rural Tanzanian district: a case for implementing a birth plan intervention. BMC Pregnancy Childbirth. 2010 Mar 19;10:13. doi: 10.1186/1471-2393-10-13. PMID 20302625
- [Result] Knol MJ, Vandenbroucke JP, Scott P, Egger M. What do case-control studies estimate? Survey of methods and assumptions in published case-control research. Am J Epidemiol. 2008 Nov 1;168(9):1073-81. doi: 10.1093/aje/kwn217. Epub 2008 Sep 15. PMID 18794220
- [Result] Mushi D, Mpembeni R, Jahn A. Effectiveness of community based Safe Motherhood promoters in improving the utilization of obstetric care. The case of Mtwara Rural District in Tanzania. BMC Pregnancy Childbirth. 2010 Apr 1;10:14. doi: 10.1186/1471-2393-10-14. PMID 20359341
- [Result] Thatte N, Mullany LC, Khatry SK, Katz J, Tielsch JM, Darmstadt GL. Traditional birth attendants in rural Nepal: knowledge, attitudes and practices about maternal and newborn health. Glob Public Health. 2009;4(6):600-17. doi: 10.1080/17441690802472406. PMID 19431006
- [Result] Kwast BE. Reduction of maternal and perinatal mortality in rural and peri-urban settings: what works? Eur J Obstet Gynecol Reprod Biol. 1996 Oct;69(1):47-53. doi: 10.1016/0301-2115(95)02535-9. PMID 8909956
- [Result] Maine D, Akalin MZ, Chakraborty J, de Francisco A, Strong M. Why did maternal mortality decline in Matlab? Stud Fam Plann. 1996 Jul-Aug;27(4):179-87. PMID 8875731
- [Result] Rodrigues L, Kirkwood BR. Case-control designs in the study of common diseases: updates on the demise of the rare disease assumption and the choice of sampling scheme for controls. Int J Epidemiol. 1990 Mar;19(1):205-13. doi: 10.1093/ije/19.1.205. PMID 2190942
- See also: http://www.uonbi.ac.ke/activities/KNHUoN — http://www.uonbi.ac.ke
- See also: http://www.popcouncil.org/pdfs/2012RH_APHIAII_CommunityMidwifery.pdf — http://www.popcouncil.org